CLINICAL TRIAL: NCT03570216
Title: Acute Effects of High-Intensity Interval Exercise vs. Moderate-Intensity Continuous Exercise on Arterial Stiffness in Chronic Stroke
Brief Title: Cardiovascular Effects of Acute Exercise Post-Stroke
Acronym: ACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ada Tang, Associate Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3113
Record Dates: First submitted 2018-03-26; First posted 2018-06-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Cardiovascular
Keywords: acute exercise; High-intensity interval exercise; feasibility; arterial stiffness
MeSH Terms: conditions — Myocardial Infarction | interventions — Exercise Test; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This will be a single group prospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): All participants will perform 3 exercise sessions: one session to assess their cardiorespiratory fitness, one session on moderate-intensity continuous exercise and one session of high-intensity interval exercise
  Interventions: Other: Cardiopulmonary exercise test; Other: Moderate-intensity continuous exercise; Other: High-intensity interval exercise

INTERVENTIONS:
Other: Cardiopulmonary exercise test — Participants will perform a graded cardiopulmonary exercise test to asses their cardiorespiratory fitness. It will also provide a peak exercise stimulus to examine acute changes in arterial stiffness, and to prescribe both moderate intensity continuous exercise and high intensity interval exercise.
Other: Moderate-intensity continuous exercise — Participants will perform a 30-minute session of moderate-intensity continuous exercise.
Other: High-intensity interval exercise — 1 week later, participants will perform a 19-minute session of high-intensity interval exercise.

SUMMARY:
There is an urgent need to reduce the impact of stroke by promoting optimal rehabilitation strategies that decrease the risk of stroke. Improving cardiovascular health following a stroke is a key rehabilitation strategy that has the potential to reduce the risk of a recurrent event.

Adverse cardiovascular events, including stroke, are often due to chronic atherosclerosis, which shows as increased arterial stiffness. Elevated arterial stiffness is prevalent in individuals with cardiovascular disease, is associated with markers of silent cerebrovascular disease and is a new marker for predicting cardiovascular risk. Cardiopulmonary exercise tests (CPETs) are used to assess cardiorespiratory fitness. Novel CPET protocols have emerged for stroke, enabling safe and valid measurements of cardiorespiratory fitness. Cardiovascular exercise, typically performed through moderate-intensity continuous exercise (MICE), can improve function and fitness in individuals living with stroke and lower the risk of recurrent stroke. Recently, high-intensity interval exercise (HIIE) has emerged as a potentially potent stimulus that may also lead to improvements in function and fitness. While HIIE has shown benefits in clinical and non-clinical populations, only a few small, preliminary studies have examined the effects of HIIE in individuals living with stroke, and most have primarily focused on examining the effects of HIIE on function and gait. No study has examined and compared the acute effects of a CPET, MICE and HIIE on arterial stiffness in stroke. This study will (1) examine the acute effects of a single session of this HIIE protocol compared to a CPET and a single session of MICE on arterial stiffness among individuals with chronic stroke, and (2) the feasibility of a high-intensity interval training exercise protocol previously found to be tolerable and effective in attaining high levels of exercise intensity in in these individuals.

DETAILED DESCRIPTION:
Stroke is the leading cause of adult disability and the fourth leading cause of death in Canada, with an annual cost to the economy of $3.6 billion. There is an urgent need to reduce the impact of stroke by promoting optimal rehabilitation strategies that decrease the risk of stroke. Improving cardiovascular health following a stroke is a key rehabilitation strategy that has the potential to reduce the risk of a recurrent event. Adverse cardiovascular events, including stroke, are often due to chronic atherosclerosis. Amplified arterial stiffness is a sign of atherosclerosis which increases arterial wall stress and reduces coronary perfusion. Elevated arterial stiffness is prevalent in individuals with cardiovascular disease, is associated with markers of silent cerebrovascular disease and is a new marker for predicting cardiovascular risk. Cardiopulmonary exercise tests (CPETs) are the gold standard for assessing cardiorespiratory fitness. In stroke, impairments in physical function may be present and limit individuals' ability to perform a CPET on traditional modes such as a cycle ergometer or treadmill. Thus, novel CPET protocols have been developed to allow individuals with stroke perform a fitness test safely and effectively. Cardiovascular exercise, typically performed through moderate-intensity continuous exercise (MICE), can improve function and fitness in individuals living with stroke and lower the risk of recurrent stroke. Recently, high-intensity interval exercise (HIIE) has emerged as a potentially potent stimulus that may also lead to improvements in function and fitness. HIIE combines short bursts of high-intensity cardiovascular exercise with periods of rest or recovery, and allows individuals to achieve higher intensities of cardiovascular exercise that do not need to be maintained for a long period of time like MICE. In this way, HIIE has the potential to be an additional exercise strategy to enhance cardiovascular health post-stroke. While HIIE has shown benefits in clinical and non-clinical populations, only a few small, preliminary studies have examined the effects of HIIE in individuals living with stroke, and most have primarily focused on examining the effects of HIIE on function and gait.

While the chronic effects of exercise on arterial stiffness have been examined in stroke, no study has examined the acute effects of a CPET, MICE, or HIIE. Different exercise stimuli may elicit variable short-term influences on arterial stiffness in individuals who have had a stroke, but this has not been previously examined. The feasibility of HIIE for individuals with a broader range of functional abilities after stroke is also not well established.

This study will (1) compare the acute effects of a HIIE session to a CPET and a session of MICE on arterial stiffness and (2) examine the feasibility of a HIIE protocol in individuals with a broad range of abilities after stroke. The investigators anticipate that (1) arterial stiffness will be elevated to a greater degree immediately following HIIE compared to the CPET and MICE, and will remain elevated following 15 minutes post-exercise, and (2) both HIIE and MICE protocols will be safe and feasible for individuals with stroke (no occurrence of adverse events), however the HIIE protocol will allow participants to obtain and be able to sustain a higher level of exercise intensity, and therefore a higher heart rate, compared to MICE. Understanding the time course of changes in arterial stiffness following acute exercise may provide insight into vascular responses of HIIE and thus potential underlying physiological mechanisms of post-stroke exercise.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age
* >6 months following first-ever, single stroke
* Living in the community (not in an institutional setting)
* Able to walk at least 10 meters (assistive devices permitted)
* Able to follow commands.

Exclusion Criteria:

* Individuals will be excluded if they present with:
* Significant disability (a score >2 in the modified Rankin scale)
* Class C or D American Heart Association Risk Scores
* Any contraindications to exercise testing or training as set forth by the American College of Sports Medicine Guidelines for Exercise Testing and Prescription (ACSM, 2014)
* Any other neurological or musculoskeletal condition or co-morbidity that would preclude safe exercise participation
* Pain worsened with exercise
* Any cognitive, communication, or behavioral concerns that could limit safe exercise involvement

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Arterial Stiffness | Resting before exercise, immediately following (within 5 minutes) of exercise cessation, and continuously for 15 minutes post exercise.
  Arterial stiffness will be measured at rest, immediately after each exercise stimulus, and continuously for 15 minutes after each exercise stimulus to assess change in this measure post-acute exercise. Arterial stiffness will be measured using the criterion standard for measuring central arterial stiffness, carotid-femoral pulse wave velocity (cfPWV). Arterial stiffness will be assessed non-invasively through applanation tonometry. cfPWV is calculated as cfPWV=D (meters)/Δt (seconds), where Δt is the pulse transit time between carotid and femoral arteries and D the distance between the two arteries.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events [Safety] | During active engagement of HIIE and MICE protocols, and within 7 days later
  Incidence of adverse events that occur during or after HIIE and MICE
Time spent at prescribed heart rate intensity [Feasibility] | During active engagement of HIIE and MICE protocols
  The total time spent at the prescribed heart rate intensity for each protocol will be determined, i.e. # minutes during the 30-minute MICE and 19- minute HIIE protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Ada Tang, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashor AW, Lara J, Siervo M, Celis-Morales C, Mathers JC. Effects of exercise modalities on arterial stiffness and wave reflection: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Oct 15;9(10):e110034. doi: 10.1371/journal.pone.0110034. eCollection 2014. PMID 25333969
- [Background] Attina TM, Drummond ID, Malatino LS, Maxwell SR, Webb DJ. Phosphodiesterase type 5 inhibition improves arterial stiffness after exercise but not exercise capacity in hypertensive men. Am J Hypertens. 2013 Mar;26(3):342-50. doi: 10.1093/ajh/hps057. Epub 2013 Jan 7. PMID 23382484
- [Background] Baert I, Daly D, Dejaeger E, Vanroy C, Vanlandewijck Y, Feys H. Evolution of cardiorespiratory fitness after stroke: a 1-year follow-up study. Influence of prestroke patients' characteristics and stroke-related factors. Arch Phys Med Rehabil. 2012 Apr;93(4):669-76. doi: 10.1016/j.apmr.2011.09.022. Epub 2012 Feb 13. PMID 22336102
- [Background] Barodka VM, Joshi BL, Berkowitz DE, Hogue CW Jr, Nyhan D. Review article: implications of vascular aging. Anesth Analg. 2011 May;112(5):1048-60. doi: 10.1213/ANE.0b013e3182147e3c. Epub 2011 Apr 7. PMID 21474663
- [Background] Ben-Shlomo Y, Spears M, Boustred C, May M, Anderson SG, Benjamin EJ, Boutouyrie P, Cameron J, Chen CH, Cruickshank JK, Hwang SJ, Lakatta EG, Laurent S, Maldonado J, Mitchell GF, Najjar SS, Newman AB, Ohishi M, Pannier B, Pereira T, Vasan RS, Shokawa T, Sutton-Tyrell K, Verbeke F, Wang KL, Webb DJ, Willum Hansen T, Zoungas S, McEniery CM, Cockcroft JR, Wilkinson IB. Aortic pulse wave velocity improves cardiovascular event prediction: an individual participant meta-analysis of prospective observational data from 17,635 subjects. J Am Coll Cardiol. 2014 Feb 25;63(7):636-646. doi: 10.1016/j.jacc.2013.09.063. Epub 2013 Nov 13. PMID 24239664
- [Background] Billinger SA, Boyne P, Coughenour E, Dunning K, Mattlage A. Does aerobic exercise and the FITT principle fit into stroke recovery? Curr Neurol Neurosci Rep. 2015;15(2):519. doi: 10.1007/s11910-014-0519-8. PMID 25475494
- [Background] Billinger SA, Coughenour E, Mackay-Lyons MJ, Ivey FM. Reduced cardiorespiratory fitness after stroke: biological consequences and exercise-induced adaptations. Stroke Res Treat. 2012;2012:959120. doi: 10.1155/2012/959120. Epub 2011 Aug 14. PMID 21876848
- [Background] Boyne P, Dunning K, Carl D, Gerson M, Khoury J, Rockwell B, Keeton G, Westover J, Williams A, McCarthy M, Kissela B. High-Intensity Interval Training and Moderate-Intensity Continuous Training in Ambulatory Chronic Stroke: Feasibility Study. Phys Ther. 2016 Oct;96(10):1533-1544. doi: 10.2522/ptj.20150277. Epub 2016 Apr 21. PMID 27103222
- [Background] Boyne P, Dunning K, Carl D, Gerson M, Khoury J, Kissela B. Within-session responses to high-intensity interval training in chronic stroke. Med Sci Sports Exerc. 2015 Mar;47(3):476-84. doi: 10.1249/MSS.0000000000000427. PMID 24977698
- [Background] Brott T, Adams HP Jr, Olinger CP, Marler JR, Barsan WG, Biller J, Spilker J, Holleran R, Eberle R, Hertzberg V, et al. Measurements of acute cerebral infarction: a clinical examination scale. Stroke. 1989 Jul;20(7):864-70. doi: 10.1161/01.str.20.7.864. PMID 2749846
- [Background] Chen Y, Shen F, Liu J, Yang GY. Arterial stiffness and stroke: de-stiffening strategy, a therapeutic target for stroke. Stroke Vasc Neurol. 2017 Mar 17;2(2):65-72. doi: 10.1136/svn-2016-000045. eCollection 2017 Jun. PMID 28959494
- [Background] Cohn JN. Arterial stiffness, vascular disease, and risk of cardiovascular events. Circulation. 2006 Feb 7;113(5):601-3. doi: 10.1161/CIRCULATIONAHA.105.600866. No abstract available. PMID 16461830
- [Background] Eng JJ, Dawson AS, Chu KS. Submaximal exercise in persons with stroke: test-retest reliability and concurrent validity with maximal oxygen consumption. Arch Phys Med Rehabil. 2004 Jan;85(1):113-8. doi: 10.1016/s0003-9993(03)00436-2. PMID 14970978
- [Background] Flansbjer UB, Holmback AM, Downham D, Patten C, Lexell J. Reliability of gait performance tests in men and women with hemiparesis after stroke. J Rehabil Med. 2005 Mar;37(2):75-82. doi: 10.1080/16501970410017215. PMID 15788341
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Gowland C, Stratford P, Ward M, Moreland J, Torresin W, Van Hullenaar S, Sanford J, Barreca S, Vanspall B, Plews N. Measuring physical impairment and disability with the Chedoke-McMaster Stroke Assessment. Stroke. 1993 Jan;24(1):58-63. doi: 10.1161/01.str.24.1.58. PMID 8418551
- [Background] Kaminsky LA, Arena R, Beckie TM, Brubaker PH, Church TS, Forman DE, Franklin BA, Gulati M, Lavie CJ, Myers J, Patel MJ, Pina IL, Weintraub WS, Williams MA; American Heart Association Advocacy Coordinating Committee, Council on Clinical Cardiology, and Council on Nutrition, Physical Activity and Metabolism. The importance of cardiorespiratory fitness in the United States: the need for a national registry: a policy statement from the American Heart Association. Circulation. 2013 Feb 5;127(5):652-62. doi: 10.1161/CIR.0b013e31827ee100. Epub 2013 Jan 7. No abstract available. PMID 23295916
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Kortianou EA, Nasis IG, Spetsioti ST, Daskalakis AM, Vogiatzis I. Effectiveness of Interval Exercise Training in Patients with COPD. Cardiopulm Phys Ther J. 2010 Sep;21(3):12-9. PMID 20957074
- [Background] Mackay-Lyons MJ, Makrides L. Exercise capacity early after stroke. Arch Phys Med Rehabil. 2002 Dec;83(12):1697-702. doi: 10.1053/apmr.2002.36395. PMID 12474172
- [Background] Mackay, J.& M.G., 2004. Atlas of Heart Disease and Stroke. Geneva: World Health Organization.,
- [Background] Madden KM, Lockhart C, Cuff D, Potter TF, Meneilly GS. Short-term aerobic exercise reduces arterial stiffness in older adults with type 2 diabetes, hypertension, and hypercholesterolemia. Diabetes Care. 2009 Aug;32(8):1531-5. doi: 10.2337/dc09-0149. Epub 2009 Jun 9. PMID 19509011
- [Background] Mattace-Raso FU, van der Cammen TJ, Hofman A, van Popele NM, Bos ML, Schalekamp MA, Asmar R, Reneman RS, Hoeks AP, Breteler MM, Witteman JC. Arterial stiffness and risk of coronary heart disease and stroke: the Rotterdam Study. Circulation. 2006 Feb 7;113(5):657-63. doi: 10.1161/CIRCULATIONAHA.105.555235. PMID 16461838
- [Background] Mohan KM, Wolfe CD, Rudd AG, Heuschmann PU, Kolominsky-Rabas PL, Grieve AP. Risk and cumulative risk of stroke recurrence: a systematic review and meta-analysis. Stroke. 2011 May;42(5):1489-94. doi: 10.1161/STROKEAHA.110.602615. Epub 2011 Mar 31. PMID 21454819
- [Background] Mutter AF, Cooke AB, Saleh O, Gomez YH, Daskalopoulou SS. A systematic review on the effect of acute aerobic exercise on arterial stiffness reveals a differential response in the upper and lower arterial segments. Hypertens Res. 2017 Feb;40(2):146-172. doi: 10.1038/hr.2016.111. Epub 2016 Oct 13. PMID 27733765
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Nichols WW, Edwards DG. Arterial elastance and wave reflection augmentation of systolic blood pressure: deleterious effects and implications for therapy. J Cardiovasc Pharmacol Ther. 2001 Jan;6(1):5-21. doi: 10.1177/107424840100600102. PMID 11452332
- [Background] Pang MY, Eng JJ, Dawson AS, McKay HA, Harris JE. A community-based fitness and mobility exercise program for older adults with chronic stroke: a randomized, controlled trial. J Am Geriatr Soc. 2005 Oct;53(10):1667-74. doi: 10.1111/j.1532-5415.2005.53521.x. PMID 16181164
- [Background] Pase MP, Beiser A, Enserro D, Xanthakis V, Aparicio H, Satizabal CL, Himali JJ, Kase CS, Vasan RS, DeCarli C, Seshadri S. Association of Ideal Cardiovascular Health With Vascular Brain Injury and Incident Dementia. Stroke. 2016 May;47(5):1201-6. doi: 10.1161/STROKEAHA.115.012608. Epub 2016 Apr 12. PMID 27073239
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362
- [Background] Rognmo O, Hetland E, Helgerud J, Hoff J, Slordahl SA. High intensity aerobic interval exercise is superior to moderate intensity exercise for increasing aerobic capacity in patients with coronary artery disease. Eur J Cardiovasc Prev Rehabil. 2004 Jun;11(3):216-22. doi: 10.1097/01.hjr.0000131677.96762.0c. PMID 15179103
- [Background] Seshadri S, Beiser A, Kelly-Hayes M, Kase CS, Au R, Kannel WB, Wolf PA. The lifetime risk of stroke: estimates from the Framingham Study. Stroke. 2006 Feb;37(2):345-50. doi: 10.1161/01.STR.0000199613.38911.b2. Epub 2006 Jan 5. PMID 16397184
- [Background] Tabara Y, Yuasa T, Oshiumi A, Kobayashi T, Miyawaki Y, Miki T, Kohara K. Effect of acute and long-term aerobic exercise on arterial stiffness in the elderly. Hypertens Res. 2007 Oct;30(10):895-902. doi: 10.1291/hypres.30.895. PMID 18049020
- [Background] Tanaka H, Dinenno FA, Monahan KD, Clevenger CM, DeSouza CA, Seals DR. Aging, habitual exercise, and dynamic arterial compliance. Circulation. 2000 Sep 12;102(11):1270-5. doi: 10.1161/01.cir.102.11.1270. PMID 10982542
- [Background] Tang A, Eng JJ, Krassioukov AV, Madden KM, Mohammadi A, Tsang MY, Tsang TS. Exercise-induced changes in cardiovascular function after stroke: a randomized controlled trial. Int J Stroke. 2014 Oct;9(7):883-9. doi: 10.1111/ijs.12156. Epub 2013 Oct 22. PMID 24148695
- [Background] Tang A, Sibley KM, Thomas SG, McIlroy WE, Brooks D. Maximal exercise test results in subacute stroke. Arch Phys Med Rehabil. 2006 Aug;87(8):1100-5. doi: 10.1016/j.apmr.2006.04.016. PMID 16876556
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Background] ACSM, 2010. ACSM's guidelines for exercise testing and prescription 8th Edition, Philadelphia: Lippincott Williams & Wilkins.